CLINICAL TRIAL: NCT03215433
Title: Single-centre, Observational Study, Concerning Blood-lipid Biomarkers of the Response to Treatment With Biotine, Prescribed in the Context of a Nominative TAU (Temporary Authorized Use) in Patients With an Inactive Progressive Form of Multiple Sclerosis (MS).
Brief Title: Study of Biomarkers of the Response to Biotine
Acronym: BIOMARBIOT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MOREAU MedDay 2016
Record Dates: First submitted 2017-06-26; First posted 2017-07-12 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis; Biotine
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biotine is proposed by neurologists to patients with a progressive form of Multiple sclerosis (MS) in the context of a nominative temporary authorization for use (TAU) as a disease-modifying treatment for their MS. A recent study showed that with this treatment, more patients experienced an improvement after one year in comparison with patients given a placebo.

The objective of this study is to identify blood biomarkers to determine good responders as early as possible. In addition, the blood parameters studied will make it possible to better understand the mechanisms of action, that have a beneficial effect on multiple sclerosis.

The management of patients will not be modified: same number of consultations (at the prescription, at 3 months, at 12 months), same clinical examination, and the same number of blood samples (at the prescription, at 3 months, and at 12 months).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* inactive progressive form of MS according to the Lublin classification and recorded in the Burgundy EDMUS database
* Patients with health insurance cover
* Patients who have provided written informed consent (OFSEP)

Exclusion Criteria:

* Patients unable to understand the information sheet
* Patients with remittent or active progressive MS
* Patients with a change in the disease-modifying treatment within the previous 3 months
* Patients treated with corticosteroids in the month before inclusion
* Impossibility to provide patients with the necessary information
* Patients in custody
* Patients under guardianship

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 25 patients with progressive (primary or secondary) MS will be encountered over time during consultations at Dijon CHU. Treatment with biotine will be proposed to patients and a nominative TAU will be requested.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
validated disability scale (EDSS) | change from baseline validated disability scale at 3 and 12 months
Walking test | change from baseline walking test at 3 and 12 months
Evolution of blood lipid biomarkers | change from baseline evolution of biomarkers at 3 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France